CLINICAL TRIAL: NCT01849120
Title: Does Near Infrared Spectroscopy Predict Low Cardiac Output State in Neonates and Infants Following Cardiac Surgery for Congenital Heart Disease?
Brief Title: NIRS Predict Low Cardiac Output State in Neonates and Infants in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Nonin Medical, Inc (Industry)
Responsible Party: Principal Investigator, William C. Oliver, William Oliver, MD, Mayo Clinic
Other Study IDs: 12-003690
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Congenital Heart Disease
Keywords: near infrared spectroscopy (NIRS); EQUANOX Advance 8004CB probes; cerebral vascular circulation; peripheral perfusion
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Near-infrared spectroscopy (NIRS): After cardiac surgery, all subjects will have EQUANOX Advance 8004CB sensors applied to peripheral sites (left and right calf and side of abdomen).
  Interventions: Device: EQUANOX Advance 8004CB sensor

INTERVENTIONS:
Device: EQUANOX Advance 8004CB sensor — The EQUANOX Advance 8004CB sensors placed in peripheral sites of neonates and infants will be used to detect peripheral perfusion and oxygen delivery.

SUMMARY:
Neonates and infants that have cardiac surgery with cardiopulmonary bypass (CPB) for congenital heart disease are at great risk for experiencing life-threatening low cardiac output syndrome (LCOS) in the first 24 hours after surgery. The poor perfusion and inadequate oxygen delivery that occurs may result in multiple organ failure and death. It is LCOS that is responsible for the majority of early postoperative deaths in this population of neonates and infants. Improved pediatric probes placed in peripheral locations using near infrared spectroscopy (NIRS) may permit continuous monitoring of venous saturations reflecting overall perfusion and oxygen balance in the tissues. Following parental or guardian consent, 30 neonates and infants scheduled to undergo surgery for congenital heart disease will be enrolled. At the end of surgery, four EQUANOX Advance 8004CB probes will be placed on the flank, lower extremities and the forehead. Continuous NIRS saturations will be monitored and stored for analysis. Point of care (POC) lactates will be obtained after admission to the intensive care unit (ICU) every 2 hours for the first 24 hours postoperatively, then once at 48 hours. The association between NIRS oxygen saturation and POC lactate values will be assessed using mixed linear models taking into account the repeated measures design. Exploratory analyses will be performed to assess whether NIRS oxygen saturation is associated with outcomes such as days in ICU, adverse events and mortality.

The ability to use noninvasive, continuous monitoring for overall perfusion and cardiac output will allow better and earlier therapy for neonates and infants following cardiac surgery.

ELIGIBILITY:
Inclusion:

* pediatric patients 0-3 years of age
* scheduled to undergo cardiopulmonary bypass surgery (CPB) for repair of congenital heart defects

Exclusion:

* weight < 2 kg or > 20 kg
* greater than 3 years of age
* thrombosed femoral arteries
* prior fasciotomies
* currently on extracorporeal membrane oxygenation (ECMO)

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric cardiac surgical patients that required cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Venous lactate level | 48 hours post surgery

SECONDARY OUTCOMES:
Blood oxygen saturation level | 48 hours after surgery
  Oxygen saturation level will be measured by near-infrared spectroscopy (NIRS).

CONTACTS AND LOCATIONS:
Overall Officials: William Oliver, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States